CLINICAL TRIAL: NCT03389152
Title: Evaluation of SWE as a Predictive Tool for Progression of Chronic Liver Diseases
Brief Title: SWE Liver Stiffness as a Predictor of Progression of Chronic Liver Diseases
Acronym: SWE Predict
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Collaborators: University of Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: LE3
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Liver Fibroses
MeSH Terms: conditions — Liver Cirrhosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Elastography — liver stiffness measurements by shear wave-based elastography

SUMMARY:
This study is a multicenter individual patient-based meta-analysis that will assess the performances of liver stiffness measurements performed with supersonic shear imaging shearwave elastography (SSI-SWE) in patients with liver fibrosis to predict progression of chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had received a liver ultrasound exam at baseline for a suspected chronic fibrotic liver disease of viral and/or steatotic origin,
* Patients who had reached the age of majority in their countries, at baseline,
* Patients with a baseline liver biopsy for histological evaluation of liver fibrosis with a length ≥ 15 mm paraffin sections (except if cirrhosis),
* Patients for whom a minimum length of clinical follow-up from baseline of 1 year had been recorded

Exclusion Criteria:

* Cause of chronic liver disease other than viral, ALD or NAFLD ( hemochromatosis, autoimmune hepatitis, biliary tract disease intrahepatic...)
* Any systemic, viral hepatitis and HIV co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed chronic liver disease of viral and/or steatotic origin, requiring a percutaneous liver biopsy, and who had received a liver ultrasound exam at baseline for a suspected chronic fibrotic liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 2148 (Actual)
Dates: Start 2007-07-26 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Liver disease progression rate | Minimum of 28 days follow-up
  Clinical signs of liver decompensation
Mortality rate | Minimum of 28 days follow-up
  Patient's death

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the study, sharing of IPD will not be required.

REFERENCES:
- [Background] Herrmann E, de Ledinghen V, Cassinotto C, Chu WC, Leung VY, Ferraioli G, Filice C, Castera L, Vilgrain V, Ronot M, Dumortier J, Guibal A, Pol S, Trebicka J, Jansen C, Strassburg C, Zheng R, Zheng J, Francque S, Vanwolleghem T, Vonghia L, Manesis EK, Zoumpoulis P, Sporea I, Thiele M, Krag A, Cohen-Bacrie C, Criton A, Gay J, Deffieux T, Friedrich-Rust M. Assessment of biopsy-proven liver fibrosis by two-dimensional shear wave elastography: An individual patient data-based meta-analysis. Hepatology. 2018 Jan;67(1):260-272. doi: 10.1002/hep.29179. Epub 2017 Nov 15. PMID 28370257
- [Derived] Gu W, de Ledinghen V, Aube C, Krag A, Strassburg C, Castera L, Dumortier J, Friedrich-Rust M, Pol S, Grgurevic I, Zeleke Y, Praktiknjo M, Schierwagen R, Klein S, Francque S, Gottfriedova H, Sporea I, Schindler P, Rennebaum F, Brol MJ, Schulz M, Uschner FE, Fischer J, Margini C, Wang W, Delamarre A, Best J, Canbay A, Bauer DJM, Simbrunner B, Semmler G, Reiberger T, Boursier J, Rasmussen DN, Vilgrain V, Guibal A, Zeuzem S, Vassord C, Vonghia L, Senkerikova R, Popescu A, Berzigotti A, Laleman W, Thiele M, Jansen C, Trebicka J. Hepatocellular Cancer Surveillance in Patients with Advanced Chronic Liver Disease. NEJM Evid. 2024 Nov;3(11):EVIDoa2400062. doi: 10.1056/EVIDoa2400062. Epub 2024 Oct 22. PMID 39437136